CLINICAL TRIAL: NCT04637672
Title: Clinical Database and Biobank of Patients With Inflammatory Myopathies: the MASC Project (Myositis, DNA, Serum, Cells) (MASC)
Acronym: MASC
Status: Completed | Type: Observational
Sponsor: Groupe Hospitalier Pitie-Salpetriere (Other)
Responsible Party: Principal Investigator, Joe Elie Salem, Clinical Professor, Groupe Hospitalier Pitie-Salpetriere
Other Study IDs: CIC-1421-20-04
Record Dates: First submitted 2020-11-08; First posted 2020-11-20 (Actual); Last update posted 2024-05-22 (Actual); Status verified 2023-09

CONDITIONS: Inflammatory Myositis; Idiopathic Inflammatory Myositis; Drug-induced Inflammatory Myositis
MeSH Terms: conditions — Myositis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 100 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Myositis are rare diseases for which the development of a cohort associated with a bank of biological samples (biobank) will allow for the conduct of researches to better delineate the underlying pathophysiology and find cures. This prospective cohort of patients with myositis will allow for identification of factors favouring the occurrence of myositis, whether they are constitutional (genetic) or acquired (environmental or drug). Different subgroups of myositis used for prognostication will be identified based on clinico-demographical variables, the nature of the organs involved beyond peripheral muscles (cardiac, diaphragm) and biomarkers abnormalities.

DETAILED DESCRIPTION:
Myositis is a rare autoimmune disease in which the immune system mistakenly attacks the patient's own peripheral muscles. This aggression manifests by muscle inflammation and necrosis responsible for a motor deficit of varying severity.

The treatments available today are insufficient and are non-specific. Biological criteria, issued from simple blood or muscle tests are missing, and they will help to define the activity of the disease and the efficacy of treatments.

The MASC protocol will include patients with myositis, and investigators will collect clinical, radiological, electrophysiological, histological and biological data to be used for researches aiming at better understanding this entity. A biobank (muscle biopsy, DNA, serum, plasma, PBMCs) will be acquired on this prospective cohort.

The study itself will be composed of a baseline visit and monthly to yearly follow-up visits which will assess:

* Clinical examination with an evaluation of the muscle strength and function impairment/handicap, including but not limited to:

  * Manual testing of proximal axial and distal muscles on the five points Medical Research Council (MRC) scale
  * Barré tests and Mingazzini tests, number of stand-up / sitting, leg crossing
* Biometry, lab and radiological measurements: muscle enzymes (creatine phosphokinase CPK, troponin, C-reactive protein, quantification of autoantibodies, muscle MRI, muscle biopsy, thorax tomodensitometry, pulmonary test function
* Extra-muscular evaluation: cardiac examination and work-up (echocardiography, cardiac MRI and Positron Emission Tomography (PET) scanner, cardiac biopsies), pulmonary evaluation, rheumatological and dermatological assessment, history of thromboembolic disease and cancer

Patient activity assessment: evaluation of daily life activity by both patient and physician using a Visual Analogue Scale

* Quality of life questionnaires
* Evaluation of the efficacy and toxicity of specific treatments

For each patient, the date of last visit or contact will be collected as well as outcomes, particularly for the cause of death if relevant.

Data from the biobank MASC " Muscles DNA/RNA Serum and Cells " will be added to other data. The biobank has been fully registered with local authorities and ethical committees ("Committee for Personal Protection (CPP)" CPP agreement). It contains peripheral blood mononuclear cells (PBMC), serum, DNA and RNA from blood and muscular biopsies collected at the diagnosis stage. The database contains immunological and genetical data.

This prospective study will also aim at:

* Identify the differential pathophysiological processes between the different subgroups of myositis
* Identify prognostic factors, including the different treatment modalities used
* Improve physiopathological knowledge (clinico-anatomobiological characteristics and identification of other biomarkers through the biobank)
* Improve the evaluation of the clinical outcomes/endpoints for future trials
* Develop clinical trials for homogeneous subgroups of patients, based on their pathophysiology and evaluated on the appropriate endpoints.

ELIGIBILITY:
Inclusion Criteria:

* All patients who had a confirmed (muscular biopsy, electromyogram, magnetic resonance imaging) or suspected clinically myositis. Myositis criteria are as follow:

  * Dermatomyositis or polymyositis according to Bohan and Peter criteria (1975)
  * Body inclusion myositis according to Griggs et al. criteria (1995)
  * Necrotizing autoimmune myopathy according to Hoogendijk et al. criteria (2004)
  * Drug-induced myositis
* Signature of the informed consent form for the study and for the biobank
* Age over 18 years old

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients who had a confirmed or suspected myositis
Sampling Method: Non-Probability Sample
Enrollment: 1273 (Actual)
Dates: Start 2013-12-19 (Actual); Primary Completion 2023-12-14 (Actual); Study Completion 2023-12-14 (Actual)

PRIMARY OUTCOMES:
Characterisation of the different myositis subgroups based on clinical, radiological, electrophysiological and histo-biological evaluations | baseline: first 30 days after inclusion
  Characterisation of the different myositis subgroups based on clinical, radiological, electrophysiological and histo-biological evaluations, including but not limited to: sexe, age, profession, a history of infection, cancer or other autoimmune and inflammatory diseases, diagnosis criteria, creatine phosphokinase, autoantibodies, immune systeme evaluation based on peripheral blood mononuclear cells, DNA sequencing muscular biopsies

SECONDARY OUTCOMES:
Characterisation of the natural history of myositis subgroups :responses to treatments, prognosis factors, evolution | up to twenty years after inclusion
  Characterisation of the natural history of myositis subgroups :responses to treatments, prognosis factors, evolution
Characterisation of an immune system signature, using peripheral blood mononuclear cells and muscular biopsies, DNA and RNA sequencing, and autoantibodies | baseline: first 30 days after inclusion
  Characterisation of an immune system signature, using peripheral blood mononuclear cells and muscular biopsies, DNA and RNA sequencing, and autoantibodies
Risk factors for All-cause mortality depending on patient's and disease characteristics | up to twenty years after inclusion
  Risk factors for All-cause mortality depending on patient's and disease characteristics including clinical, radiological electrophysiological, histo-biological and immunological as well as treatment received stratified by each subgroup of myositis
Change of the quality of life, using quality of life questionnaires, depending of patients and disease characteristics | up to twenty years after inclusion
  Change of the quality of life, using quality of life questionnaires, depending of patients and disease characteristics
Change of activity impairment using an evaluation of daily life activity by both patient and physician using a Visual Analogue Scale depending of patients and disease characteristics | up to twenty years after inclusion
  Change of activity impairment using an evaluation of daily life activity by both patient and physician using a Visual Analogue Scale depending of patients and disease characteristics
Characterisation of a quality-of-life scale using biological data (CPK), muscle weakness (muscle testing) and other visceral involvements | up to twenty years after inclusion
  Characterisation of a quality-of-life scale using biological data (CPK), muscle weakness (muscle testing) and other visceral involvements
Characterisation of a global activity scale using biological data (CPK), muscle weakness (muscle testing) and other visceral involvements | up to twenty years after inclusion
  Characterisation of a global activity scale using biological data (CPK), muscle weakness (muscle testing) and other visceral involvements
Incidence of major cardio-vascular events | up to twenty years after inclusion
  Incidence of major cardio-vascular events
Consequences on outcomes of major cardio-vascular events | up to twenty years after inclusion
  Consequences on outcomes of major cardio-vascular events
Correlation of myositis with the development of extra-muscular diseases including but not limited to dermatological, rheumatological, cardiological and pneumological associated diseases | up to twenty years after inclusion
  Correlation of myositis with the development of extra-muscular diseases including but not limited to dermatological, rheumatological, cardiological and pneumological associated diseases
Characterisation of respiratory function with pulmonary function test and thoracic tomodensitometry | up to twenty years after inclusion
  Characterisation of respiratory function with pulmonary function test and thoracic tomodensitometry
Characterisation of diaphragmatic failure with pulmonary function test and thoracic tomodensitometry | up to twenty years after inclusion
  Characterisation of diaphragmatic failure with pulmonary function test and thoracic tomodensitometry
Follow up of respiratory function with pulmonary function test and thoracic tomodensitometry | up to twenty years after inclusion
  Follow up of respiratory function with pulmonary function test and thoracic tomodensitometry
Follow up of diaphragmatic failure with pulmonary function test and thoracic tomodensitometry | up to twenty years after inclusion
  Follow up of diaphragmatic failure with pulmonary function test and thoracic tomodensitometry

CONTACTS AND LOCATIONS:
Overall Officials: Olivier Benveniste, PU PH, Study Director — Groupe Hospitalier Pitie-Salpetriere; Yves Allenbach, Study Director — Groupe Hospitalier Pitie-Salpetriere; Joe Elie SALEM, Study Director — Groupe Hospitalier Pitie-Salpetriere
Locations (1):
- AP-HP, Pitié-Salpêtrière Hospital, Department of Internal Medicine and clinical immunology, Paris, France

REFERENCES:
- [Derived] Teboul A, Allenbach Y, Tubach F, Belin L, Cassius C, Demortier J, Dossier A, Faucon C, Kasser C, Mekinian A, Monseau G, Fouchard M, Chambrelan E, Viguier M, Kluger N, Mahevas T, Bergeret B, Bachmeyer C, Lenormand C, Hotz C, Diaz E, Cordel N, Benveniste O, Bessis D, Bouaziz JD, Chasset F. Prognostic factors for patients with cancer-associated dermatomyositis: a retrospective, multicentre cohort study of 73 patients. Rheumatology (Oxford). 2025 May 1;64(5):2970-2978. doi: 10.1093/rheumatology/keae629. PMID 39589730
- [Derived] Demortier J, Vautier M, Chosidow O, Gallay L, Bessis D, Berezne A, Cordel N, Schmidt J, Smail A, Duffau P, Jachiet M, Begon E, Gottlieb J, Chasset F, Graveleau J, Marque M, Cesbron E, Forestier A, Josse S, Kluger N, Beauchene C, Le Corre Y, Pagis V, Rigolet A, Guillaume-Jugnot P, Authier FJ, Guilain N, Streichenberger N, Leonard-Louis S, Boussouar S, Landon-Cardinal O, Benveniste O, Allenbach Y. Anti-SAE autoantibody in dermatomyositis: original comparative study and review of the literature. Rheumatology (Oxford). 2023 Dec 1;62(12):3932-3939. doi: 10.1093/rheumatology/kead154. PMID 37010495